CLINICAL TRIAL: NCT01159314
Title: Baerveldt Plate Area Comparison (BPAC)
Acronym: BPAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00037146
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma
Keywords: glaucoma; Baerveldt Implants
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Baerveldt 250 mm2 (Experimental): Patients receiving Baerveldt 250 mm2
  Interventions: Procedure: Baerveldt Device surgical Procedure
- Arm B - Baerveldt 350 mm2 (Experimental): Patients receiving Baerveldt 350 mm2
  Interventions: Procedure: Baerveldt Device surgical Procedure

INTERVENTIONS:
Procedure: Baerveldt Device surgical Procedure — Implant surgery

SUMMARY:
This research is being done to compare the safety and effectiveness of two sizes of the Baerveldt glaucoma implant.

A Baerveldt glaucoma implant is one of the most common types of glaucoma operations performed. This procedure works by providing a route by which fluid can drain out of the eye to decrease the intraocular pressure. The Baerveldt implant does this by placing a tube into the eye which shunts aqueous fluid to a silicone plate which is attached to the sclera (white portion of the eye). It is this plate that comes in two different sizes (250 square millimeters and 350 square millimeters).

Earlier studies have shown that larger plate sizes produce lower eye pressures but that they may also result in more complications. While both Baerveldt devices are currently in use and have been shown to be safe and effective, it is unclear if one is superior to the other. The purpose of this study is to see if one size of device works better with fewer complications.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Intra-Ocular Pressure (IOP) > 18 mm Hg and < 40 mm Hg on medical therapy
* Previous ocular surgery limited to (cataract, corneal transplant, trabeculectomy, vitrectomy)
* Consent signed

Exclusion Criteria:

* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits
* Pregnant or nursing
* Neuro-Linguistic Programming (NLP) vision
* Iris neovascularization or proliferative retinopathy
* Epithelial or fibrous downgrowth
* Chronic or recurrent uveitis
* Steroid-induced glaucoma
* Severe posterior blepharitis
* Previous cyclodestructive procedure
* Conjunctival scarring from prior ocular trauma or cicatrizing disease (e.g. Stevens Johnson syndrome, ocular pemphigoid) precluding Baerveldt implantation.
* Functionally significant cataract
* Need for Baerveldt implant combined with other ocular procedures (ie cataract surgery,penetrating keratoplasty, or retinal surgery) or anticipated need for additional ocular surgery
* Prior glaucoma drainage device (tube) implant
* Prior retinal surgery with remaining silicone oil
* Prior scleral buckling procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-06; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Visual Acuity as assessed by Early Treatment Diabetic Retinopathy Study (EDTRS) | Up to 5 years
  Visual acuity is an important outcome variable in the BPAC. Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing will be employed at the Qualifying Assessment and at every follow-up visit.The patient starts are the top of the chart and begins to read down the chart. The patient reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified. ETDRS visual acuity is required at the Qualifying Assessment and at the 1 year, 3 year, and 5 year follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boland, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - University of California - Davis, Sacramento, California
  - U. Miami/Bascom Palmer, Miami, Florida
  - The Wilmer Eye Institute, Baltimore, Maryland
  - Mount Sinai School of Medicine, New York, New York
  - Wills Eye Institute, Philadelphia, Pennsylvania